CLINICAL TRIAL: NCT06834126
Title: DINOMITE (Decreasing Hypoxia With Mitochondrial Inhibition in Locally Advanced Rectal Cancer): Phase 1 Trial of Papaverine in Combination With Radiation
Brief Title: Papaverine in Combination With Radiation Therapy for the Treatment of Locally Advanced Rectal Cancer, DINOMITE Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24405; NCI-2024-10075 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24405 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01CA297752 (NIH)
Record Dates: First submitted 2024-12-27; First posted 2025-02-19 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Rectal Adenocarcinoma; Stage II Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — Specimen Handling; Consolidation Chemotherapy; Endoscopy, Gastrointestinal; Magnetic Resonance Spectroscopy; Papaverine; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (RT, CC) (Active Comparator): Patients undergo RT QD on days 1-5 (Monday-Friday) of week 1. Starting at week 5, patients receive SOC CC with either mFOLFOX6 or CAPOX for 3-4 months in the absence of disease progression or unacceptable toxicity. As early as four weeks following completion of CC, patients with persistent disease (non-cCR) or disease recurrence in the rectum during disease evaluation may undergo ToME. Additionally, patients undergo one fMRI on study as well as CT, MRI, endoscopy, and blood and tissue sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Consolidation Therapy; Procedure: Functional Magnetic Resonance Imaging; Procedure: Gastrointestinal Endoscopy; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Procedure: Total Mesorectal Excision
- Cohort 2 (PPV, RT, CC) (Experimental): Patients receive PPV IV over 15-30 minutes on day -3 of week 0 and days 1-5 of week 1. Patients also undergo RT QD on days 1-5 (Monday-Friday) of week 1, 1-2 hours after PPV. Starting at week 5, patients receive SOC CC with either mFOLFOX6 or CAPOX for 3-4 months in the absence of disease progression or unacceptable toxicity. As early as four weeks following completion of CC, patients with persistent disease (non-cCR) or disease recurrence in the rectum during disease evaluation may undergo ToME. Additionally, patients undergo two fMRI on study as well as CT, MRI, endoscopy, and blood and tissue sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Consolidation Therapy; Procedure: Functional Magnetic Resonance Imaging; Procedure: Gastrointestinal Endoscopy; Procedure: Magnetic Resonance Imaging; Drug: Papaverine; Radiation: Radiation Therapy; Procedure: Total Mesorectal Excision

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Consolidation Therapy — Receive CC with mFOLFOX6 or CAPOX
  Other Names: Consolidation; intensification therapy; Post Remission Therapy; Postremission Therapy
Procedure: Functional Magnetic Resonance Imaging — Undergo fMRI
  Other Names: fMRI; Functional MRI
Procedure: Gastrointestinal Endoscopy — Undergo endoscopy
  Other Names: Enteroscopy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Papaverine — Given IV
  Other Names: Cerebid; Cerespan; Pavabid; Pavacap; Pavatym; Robaxapap
  Arms: Cohort 2 (PPV, RT, CC)
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Total Mesorectal Excision — Undergo ToME
  Other Names: TME

SUMMARY:
This phase I trial studies the side effects and best dose of papaverine (PPV) when given together with radiation therapy (RT) and tests how well it works in treating patients with rectal cancer that has spread to nearby tissue or lymph nodes (locally advanced). PPV is an enzyme inhibitor, and it may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. RT uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Giving PPV with RT may be safe, tolerable, and/or effective in treating patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of papaverine (PPV) in combination with radiation therapy (RT) for locally advanced rectal cancer (LARC).

II. Describe the safety and tolerability of PPV in combination with standard of care (SOC) RT for LARC.

SECONDARY OBJECTIVES:

I. Determine the clinical complete response rate (cCR), and local-regional control rate of PPV in combination with RT for LARC.

II. Determine the total mesorectal excision (ToME)-free survival, local-regional recurrence free survival (LRRFS), disease-free survival (DFS), distant-metastasis-free survival (DMFS) and overall survival (OS) of PPV in combination with RT for LARC.

EXPLORATORY OBJECTIVES:

I. Determine whether PPV in combination with RT for LARC directly results in reduced tumor hypoxia.

II. Explore whether RT with and without mitochondrial oxygen consumption (MOC) inhibition alters the tumor immune microenvironment (TIME) in patients receiving SOC RT for LARC.

III. Explore whether molecular profiling (changes in hypoxia-induced gene expression, immune cell tumor infiltrates and peripheral immune profiling) can predict which patients may respond best to PPV in combination with SOC RT for LARC.

IV. Explore whether stool microbial signatures are associated with response to or progression after PPV in combination with SOC RT for LARC.

OUTLINE: This is a dose escalation study of PPV in combination with RT followed by a dose-expansion study. Patients are randomized to 1 of 2 cohorts.

COHORT 1: Patients undergo RT once daily (QD) on days 1-5 (Monday-Friday) of week 1. Starting at week 5, patients receive SOC consolidation chemotherapy (CC) with either modified leucovorin, fluorouracil, oxaliplatin-6 (mFOLFOX6) or capecitabine-oxaliplatin (CAPOX) for 3-4 months in the absence of disease progression or unacceptable toxicity. As early as four weeks following completion of CC, patients with persistent disease (non-cCR) or disease recurrence in the rectum during disease evaluation may undergo ToME. Additionally, patients undergo one functional magnetic resonance imaging (fMRI) on study as well as computed tomography (CT), magnetic resonance imaging (MRI), endoscopy, and blood and tissue sample collection throughout the trial.

COHORT 2: Patients receive PPV intravenously (IV) over 15-30 minutes on day -3 of week 0 and days 1-5 of week 1. Patients also undergo RT QD on days 1-5 (Monday-Friday) of week 1, 1-2 hours after PPV. Starting at week 5, patients receive SOC CC with either mFOLFOX6 or CAPOX for 3-4 months in the absence of disease progression or unacceptable toxicity. As early as four weeks following completion of CC, patients with persistent disease (non-cCR) or disease recurrence in the rectum during disease evaluation may undergo ToME. Additionally, patients undergo two fMRI on study as well as CT, MRI, endoscopy, and blood and tissue sample collection throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for an additional 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Willingness to participate in all correlative studies: fMRI, and tissue collection of tumor and normal rectum (ribonucleic acid [RNA]/deoxyribonucleic acid [DNA]/protein), blood (plasma/peripheral blood mononuclear cell [PBMC]) draws and stool collection
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed rectal adenocarcinoma
* Patient wants to pursue an organ preservation/non-operative management (NOM) approach after completion of total neoadjuvant therapy (TNT)
* Locally advanced rectal cancer (T3-4 or node+, M0)
* Tumor is microsatellite stable (MSS) (defined as not microsatellite instability-high [MSI-H] or mismatch repair deficient [dMMR])
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3 (within 30 days of start). NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets ≥ 100,000/mm^3 (within 30 days of start). NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin ≥ 9g/dL (within 30 days of start). NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (within 30 days of start)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (within 30 days of start)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (within 30 days of start)
* Creatinine clearance of ≥ 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 30 days of start)
* For patients with known infections only: seropositive for HIV, hepatitis C virus (HCV) or hepatitis B virus (HBV), nucleic acid quantitation must be performed. Viral load must be undetectable. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial (within 28 days of start)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (within 30 days of start)
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chemotherapy, biological therapy, immunotherapy within 14 days or five half-lives (whichever is shorter) prior to day 1 of protocol therapy
* Prior pelvic irradiation resulting in overlapping fields
* Use of levodopa in the last 30 days
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Unable to undergo MRI and endoscopic procedures
* History of complete atrioventricular block, hepatic dysfunction (e.g. cirrhosis), or priapism
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-09-19 (Estimated); Study Completion 2028-09-19 (Estimated)

PRIMARY OUTCOMES:
Acute dose limiting toxicity (DLT) | From time of single-agent papaverine (PPV) week 0 treatment to start of consolidation chemotherapy (CC), assessed up to 4 weeks
  As assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. A defined adverse event considered to be possibly, probably, or definitely related to study treatment (radiation therapy or PPV). Will employ the time-to-event Bayesian optimal interval design (TITE-BOIN) to find the maximum tolerated dose (MTD).
Late DLT | From the start of CC week 5 treatment to 12 months from week 0
  As assessed by NCI CTCAE v5.0. A defined adverse event considered to be possibly, probably, or definitely related to study treatment (radiation therapy or PPV). Will employ the TITE-BOIN design to find the MTD.
Incidence of treatment related adverse events during acute DLT period | From time of single-agent PPV week 0 treatment to start of CC, assessed up to 4 weeks
  As assessed by NCI CTCAE v5.0. Will be delineated by grade and attribution. A defined adverse event considered to be possibly, probably, or definitely related to study treatment (radiation therapy or PPV).
Incidence of treatment related adverse events during late DLT period | From the start of CC week 5 treatment to 12 months from week 0
  As assessed by NCI CTCAE v5.0. Will be delineated by grade and attribution. A defined adverse event considered to be possibly, probably, or definitely related to study treatment (radiation therapy or PPV).

SECONDARY OUTCOMES:
Clinical complete response rate | From time of single agent papaverine (PPV) week 0 treatment to completion of consolidation chemotherapy (CC), assessed up to 20 weeks.
  Will be defined as percent of evaluable patients having no evidence of disease as assessed by magnetic resonance imaging/endoscopy. Will be summarized by cohort and dose level.
Local-regional control rate | From time of single agent papaverine (PPV) week 0 treatment to completion of consolidation chemotherapy (CC), assessed up to 20 weeks.
  Will be defined as percent of evaluable patients having no evidence of pelvic recurrence in the areas of the primary tumor and regional lymph nodes.
Local-regional recurrence free survival | From enrollment to date of first local regional recurrence, death as a result of any cause or being censored at last contact, assessed up to 5 years
Total mesorectal excision free survival | From enrollment to date of total mesorectal surgical excision, death as result of any cause or being censored at last contact, assessed up to 5 years
Disease-free survival | From enrollment to date of first disease recurrence, death as a result of any cause or being censored at last contact, assessed up to 5 years
Distant-metastasis-free survival | From enrollment to date of first distant metastases occurrence, death as a result of any cause or being censored at last contact, assessed up to 5 years
Overall survival | From enrollment to date of death as a result of any cause or being censored at last contact, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Terence M Williams, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States